CLINICAL TRIAL: NCT05811962
Title: The Role of Serum Amyloid A in Clinical Decision-making Concerning Sarcoidosis Patients
Brief Title: The Diagnostic and Prognostic Role of SAA in Intrathoracic Sarcoidosis
Acronym: SARCO
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Zala Leštan, Principal Investigator, University Medical Centre Ljubljana
Other Study IDs: UMCLjubljanaPulmo
Record Dates: First submitted 2023-03-16; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: Sarcoidosis, Pulmonary
MeSH Terms: conditions — Sarcoidosis, Pulmonary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum samples for biomarker analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intrathoracic sarcoidosis cohort: Patients with intrathoracic sarcoidosis, confirmed according to European Respiratory Society/ World Association of Sarcoidosis and Other Granulomatous disease (ERS/WASOG) criteria
  Interventions: Other: No intervention
- Healthy controls: Healthy blood donors

INTERVENTIONS:
Other: No intervention — No intervention, only comparison
  Groups: Intrathoracic sarcoidosis cohort

SUMMARY:
The goal of this observational study is to elucidate the role of serum amyloid A (SAA) in the diagnosis and follow-up of sarcoidosis, including its prognostic value. The main questions it aims to answer are:

* Whether, at the time of diagnosis, SAA is in correlation with other serum markers of granulomatous inflammation, interstitial disease and pulmonary fibrosis, lung function and radiologic characteristics of intrathoracic sarcoidosis,
* Whether increased serum concentrations of SAA at the time of diagnosis act as a prognostic marker of progressive granulomatous inflammation and pulmonary interstitial disease.

Patients will undergo standard diagnostic procedures for intrathoracic sarcoidosis, according to WASOG (World association of sarcoidosis and other granulomatous disorders) criteria. Two additional vials of blood will be taken at diagnosis and one vial at follow-up for serum processing and biomarker analysis.

Healthy blood donors will represent our group of healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years of age
* Enrolled immediately after the first diagnostic workup and before any treatment was initiated.

Exclusion Criteria:

* Individuals with granulomatous disease that could not be unequivocally diagnosed as sarcoidosis were excluded, as well as patients with possible confounding other known systemic inflammatory illnesses, acute infection, patients on immunosuppressive drugs or immunotherapy and patients with active cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * All patients comply with the accepted European Respiratory Society/ World Association of Sarcoidosis and Other Granulomatous disease (ERS/WASOG) guidelines for the diagnosis of sarcoidosis and have undergone complete functional and radiological assessment, including spirometry.
  * Histological confirmation of non-caseating granulomas in thoracic lymph nodes and lung parenchyma has been obtained by flexible bronchoscopy, as well as bronchoalveolar lavage (BAL) fluid for the determination of BAL CD4+/CD8+ ratio.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
The correlation of mean serum concentration of serum amyloid A (SAA) in patients, newly diagnosed with intrathoracic sarcoidosis to mean value in healthy controls | 4 years for patient enrollment
  The mean serum concentration of serum amyloid A (SAA) (in micrograms per millilitre) in patients, newly diagnosed with intrathoracic sarcoidosis will be determined for our entire intrathoracic sarcoidosis cohort and separately first for patients in different Scadding stages (0-4) and secondly according to high-resolution computed tomography (HRCT) pattern (lymph node enlargement, peribronchovascular/perilymphatic lesions, ground-glass lesions and pulmonary fibrosis). The mean values will then be compared to the mean value of SAA in healthy controls to determine possible statistically significant differences.
The correlation of serum concentrations of serum amyloid A (SAA) at the time of diagnosis of intrathoracic sarcoidosis with serum concentrations of other biomarkers of granulomatous inflammation and pulmonary interstitial disease. | 4 years for patient enrollment
  We will determine whether serum concentrations of SAA at the time of diagnosis of intrathoracic sarcoidosis corelate to serum concentrations of granulomatous disease markers (CC chemokine ligand 18 (CCL18), monokine induced by interferon-γ (CXCL9), interferon-γ-induced protein 10 (CXCL10)) and activity of serum chitotriosidase (CTO) and serum concentrations of biomarkers of interstitial lung disease and lung fibrosis (surfactant protein D (SP-D) and cancer antigen 15.3 (CA 15.3)/Krebs von den Lungen 6 (KL-6)).
Correlation of serum concentrations of SAA at the time of diagnosis of intrathoracic sarcoidosis to pulmonary function test results. | 4 years for patient enrollment
  We will determine whether serum concentrations of SAA corelate to results of lung function tests (percentages predicted of forced vital capacity, forced expiratory volume in 1 second and diffusion capacity for carbon monoxide) at the time of diagnosis of intrathoracic sarcoidosis.
Correlation of serum concentrations of SAA at the time of diagnosis of intrathoracic sarcoidosis to radiologic extent of disease. | 4 years for patient enrollment
  We will determine whether serum concentrations of SAA at the time of diagnosis of intrathoracic sarcoidosis correlate with extent of disease on HRCT, expressed in percentage of pulmonary parenchyma involved (0%, 0-33%, 33-66%, 66-100%).
Correlation of serum concentrations of SAA at the time of diagnosis of intrathoracic sarcoidosis to changes in lung function tests after 3 years of follow-up. | 3 years follow-up
  We will determine whether SAA concentrations at the time of diagnosis of intrathoracic sarcoidosis correlate with changes in lung function tests (percentages predicted of forced vital capacity, forced expiratory volume in 1 second and diffusion capacity for carbon monoxide) at patient follow-up after 3 years.
Correlations of serum concentrations of SAA at the time of diagnosis of intrathoracic sarcoidosis to changes in HRCT disease extent after 3 years of follow-up. | 3 years follow-up
  We will determine whether SAA concentrations at the time of diagnosis of intrathoracic sarcoidosis correlate with changes in HRCT disease extent (descriptive terms used: resolution, stagnation, progression) at patient follow-up after 3 years.
Correlation of serum concentrations of SAA at the time of diagnosis of intrathoracic sarcoidosis to need for recent/ongoing therapy after 3 years of follow-up. | 3 years follow-up
  We will determine whether serum concentrations of SAA at the time of diagnosis of intrathoracic sarcoidosis correlate with the need for recent/ongoing therapy in patients, assessed at a 3-year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Zala Leštan Ramovš, MD, Principal Investigator — UMC Ljubljana
Locations (1):
- Department of pulmonary diseases and allergy, UMC Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iannuzzi MC, Rybicki BA, Teirstein AS. Sarcoidosis. N Engl J Med. 2007 Nov 22;357(21):2153-65. doi: 10.1056/NEJMra071714. No abstract available. PMID 18032765
- [Background] Chen ES, Song Z, Willett MH, Heine S, Yung RC, Liu MC, Groshong SD, Zhang Y, Tuder RM, Moller DR. Serum amyloid A regulates granulomatous inflammation in sarcoidosis through Toll-like receptor-2. Am J Respir Crit Care Med. 2010 Feb 15;181(4):360-73. doi: 10.1164/rccm.200905-0696OC. Epub 2009 Nov 12. PMID 19910611
- [Background] Zhou ER, Arce S. Key Players and Biomarkers of the Adaptive Immune System in the Pathogenesis of Sarcoidosis. Int J Mol Sci. 2020 Oct 7;21(19):7398. doi: 10.3390/ijms21197398. PMID 33036432
- [Background] Kraaijvanger R, Janssen Bonas M, Vorselaars ADM, Veltkamp M. Biomarkers in the Diagnosis and Prognosis of Sarcoidosis: Current Use and Future Prospects. Front Immunol. 2020 Jul 14;11:1443. doi: 10.3389/fimmu.2020.01443. eCollection 2020. PMID 32760396